CLINICAL TRIAL: NCT07276646
Title: Perioperative Opioid-sparing Effect of Retrosuperior Costotransverse Ligament Block Versus Erector Spinae Block in Laparoscopic Cholecystectomy: A Randomized Clinical Trial.
Brief Title: Perioperative Opioid-sparing Effect of Retrosuperior Costotransverse Ligament Block Versus Erector Spinae Block in Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1783
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Perioperative Analgesia
Keywords: retrosuperior costotransverse ligament block; erector spinae block; laparoscopic cholecystectomy

STUDY DESIGN:
Intervention Model Description: Achievement of high-quality perioperative opioid-sparing effect and postoperative analgesia for laparoscopic cholecystectomy with optimum hemodynamic stability and high patient and surgeon satisfaction by comparing retrosuperior costotransverse ligament block and erector spinae block in laparoscopic cholecystectomy
Who Masked: Participant, Outcomes Assessor
Masking Description: anesthesiologist not sharing in the study will assess outcomes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrosuperior costotransverse ligament block group (Active Comparator): The patient will receive retrosuperior costotransverse ligament block
  Interventions: Procedure: Retrosuperior costotransverse ligament block group
- Erector spinae block group (Active Comparator): The patient will receive erector spinae block.
  Interventions: Procedure: Erector spinae block group

INTERVENTIONS:
Procedure: Retrosuperior costotransverse ligament block group — The patient will receive retrosuperior costotransverse ligament block
  Arms: Retrosuperior costotransverse ligament block group
Procedure: Erector spinae block group — The patient will receive erector spinae block.
  Arms: Erector spinae block group

SUMMARY:
This study aims to compare the analgesic effect of retro superior costotransverse ligament space block vs erector spinae plane block to Achieve high-quality perioperative opioid-sparing effect and postoperative analgesia after laparoscopic cholecystectomy with optimum hemodynamic stability and high patient and surgeon satisfaction

DETAILED DESCRIPTION:
This study aims to compare between retro superior costotransverse ligament space block vs erector spinae plane block

* To compare the analgesic outcomes (time to first analgesic request, total amount of analgesic consumption and pain scores by NRS)
* To assess the block performance time required to perform each technique .
* To compare intraoperative parameters (hemodynamics and intraoperative fentanyl consumption)
* To assess patient, surgeon satisfaction and complications of the block.

ELIGIBILITY:
Inclusion Criteria:

1. patient acceptance
2. Age: 21-64 years old.
3. Sex: both sexes.
4. Physical status: ASA I & II.
5. Body mass index (BMI): 18.5 - 30 kg/m2.
6. Type of operations: elective laparoscopic cholecystectomy.
7. Duration of surgery not more than 2 hours.

Exclusion Criteria:

1. Known hypersensitivity to lidocaine or bupivacaine.
2. Patients with respiratory insufficiency.
3. Coagulation disorders or taking drugs affect surgical hemostasis.

7. Patients with pre-existing neurological deficits. 8. Uncooperative patient or with altered mental status. 9. Patient with advanced cardiovascular or respiratory diseases

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
The time to first call to rescue analgesia | 24 hours
  The time to first call to rescue analgesia( the interval between the block injection till the NRS more than or equal 4) (naluphine) will be recorded

SECONDARY OUTCOMES:
To assess block characteristics (block performance time) | 1 hour
  To assess block characteristics (block performance time) in minutes
Total intraoperative fentanyl consumption | duration of surgery (up to 2 hours)
  Total intraoperative fentanyl required other than the induction dose in micrograms
Pain intensity by Numerical Rating Scale | 30 minutes after arrival to post anesthesia care unit , 2hours, 4hours, 6hours, 8hours, 12hours, 18 hours and 24hours postoperative
  Analgesic parameters (Pain intensity at rest and at movement) by using Numerical Rating Scale (NRS) which will explained to patient as follows:0=no pain and 10= worst pain
total amount of rescue analgesia | 24 hours
  total amount of rescue analgesia if NRS≥4. in the first 24 hours.
Intraoperative hemodynamics (Heart Rate and Mean Arterial Pressure) | every 5 minutes in the first 30 minutes then every 10 minutes till the end of surgery
  Intraoperative hemodynamics every 5 minutes in the first 30 minutes then every 10 minutes till the end of surgery
Patient's satisfaction | 24 hours
  all patient's satisfaction: The patients will be asked to rate the overall degree of satisfaction of the analgesia by using a 5-points likert-like verbal scale (1 = very dissatisfied analgesia, 2 = dissatisfied analgesia, and 3 = neutral, 4=satisfied analgesia, and 5=very satisfied analgesia)
complication of the block | 24 hours
  complication of the block( heamatoma,local anesthetic toxicity,infection)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of human medicine, Zagazig university, Zagazig, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No